CLINICAL TRIAL: NCT05065437
Title: Immersive Virtual Reality and Noninvasive Spinal Stimulation to Promote Arm Function in Individuals With Tetraplegia
Brief Title: Virtual Reality and Spinal Stimulation to Improve Arm Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No IRB application has been prepared for this study and other studies have taken priority. The study team will not be working on this study for the foreseeable future.
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP00015240
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Tetraplegia
Keywords: upper limb function; virtual reality; spinal cord stimulation
MeSH Terms: conditions — Quadriplegia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality and spinal stimulation (Experimental): Safety and feasibility of a virtual reality and spinal stimulation intervention will be tested.
  Interventions: Other: Active (Virtual reality and spinal stimulation)

INTERVENTIONS:
Other: Active (Virtual reality and spinal stimulation) — Each session is 25 minutes; 5 minutes of setup, and 20 minutes of simultaneous spinal stimulation at the cervical level and immersive virtual experience/gameplay.

SUMMARY:
The main objective of our work is to develop and test the safety and feasibility of a home-based upper limb rehabilitation program for individuals with tetraplegia. The program will consist of simultaneous non-invasive spinal cord stimulation and immersive virtual exercises of the upper limbs, with a focus on shoulder and elbow function.

ELIGIBILITY:
Inclusion Criteria:

1. incomplete low tetraplegia (C5-8; [ASIA] classification B-D),
2. free of contraindications to transspinal stimulation,
3. more than one-year post-injury,
4. stable medication regimen for the past month,
5. utilization of wheelchair as a primary mode of mobility (>75% of the time). -

Exclusion Criteria:

1. Neurologic injury other than spinal cord injury
2. severe medical illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in medical status | Baseline to post intervention, approximately 4 weeks
  Safety of the intervention will be assessed as the number of participants who experience a reduction in medical stability and/or functionality from before to after the intervention.
Acceptability of the treatment | Post intervention, approximately 4 weeks
  Acceptability of the treatment will be assessed using the Treatment Evaluation Inventory-Short Form. Items are scored using a 5-point scale, with 1 equaling strongly disagree and 5 equaling strongly agree. TEI-SF scores can range from 9 to 45, with higher scores representing greater acceptance of the treatment.
Usability of the treatment | Post intervention, approximately 4 weeks
  Usability of the treatment will be assessed using the Usefulness, Satisfaction, and Ease of Use (USE) Questionnaire. Items are rated on a seven-point scale ranging from strongly disagree to strongly agree. A higher scale score indicates higher usability.

SECONDARY OUTCOMES:
Change in affect | Baseline to post intervention, approximately 4 weeks
  Affect will be assessed using the Positive and Negative Affect Schedule (PANAS). The PANAS is a 20-item measure that measures the intensity of 20 emotions on a 0-5 scale ranging from "not at all" to "extremely."
Change in current pain intensity | Baseline to post intervention, approximately 4 weeks
  Current pain intensity will be assessed using a Numeric Rating Scale (NRS). Participants will rate their current pain (multiple types of pain) on a 0-10 scale (0 = "no pain" and 10 = "worst possible pain").
Change in clinical muscle strength | Baseline to post intervention, approximately 4 weeks
  Clinical muscle strength will be assessed using the American Spinal Cord Injury Association (ASIA) Upper Extremity Motor Score. Motor strength is rated on a 6 point scale with higher ratings indicating greater strength.
Change in upper limb function | Baseline to post intervention, approximately 4 weeks
  Upper limb function will be assessed using the Spinal Cord Independence Measure (SCIM). The SCIM is composed of 19 items that assess function. SCIM scores range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Peterson, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No